CLINICAL TRIAL: NCT03494491
Title: Characterization of Chitin-glucan Fiber Fermentation in Human After a Single Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Nathalie Delzenne, Professor, Université Catholique de Louvain
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FiberTAG1
Record Dates: First submitted 2018-03-06; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — carboxymethyl-chitin-glucan; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Chitin-glucan — Second test day (D2), subjects will received 4.5g of chitine-glucan
Dietary Supplement: Maltodextrin — First test day (D0), subjects will received 4.5g of maltodextrin.

SUMMARY:
The aim of this research study is to characterize the fermentation of chitin-glucan fiber by assessing the volatile compounds released in the breath. For this purpose, an interventional study with control will be performed. After a single administration of 4.5 g of chitin-glucan fiber, the kinetic of production of exhaled volatile compounds (such as H2, methane, SCFAs,…) will be measured during twelve hours. These results will be compared to the exhaled volatile compounds measured during twelve hours after supplementation with 4.5g of maltodextrin (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Woman or man, aged of 18 to 40 years
* Body mass index (BMI) between 18 and 25 kg/m2
* In good general health as evidenced by medical history and physical examination
* Non-smoker
* Caucasian
* For women: use of highly effective contraception
* H2 - producer as evidenced by the screening test (described in latter section)
* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Subjects presenting gastro-intestinal disorders such as ulcers, diverticulitis and inflammatory bowel diseases
* Subject presenting allergy or food intolerance (lactose, gluten,…)
* Subjects with psychiatric problems and/or using antipsychotics
* Current or recent (< 4 weeks) intake of antibiotics, probiotics, prebiotics, fiber supplement, and/or any products modulating gut transit
* Feeding particular diet such as vegetarian diet or hyper protein diet
* Chronic intake of drug, excepted contraceptive drug
* Pregnant or lactating woman or woman who did not use highly effective contraception
* Subjects who drink more than 3 glasses of alcohol per day (> 30 g of alcohol per day)
* Subjects having participated to another clinical trial 1 month before the screening test visit
* Subjects presenting an allergy or intolerance to one component of the product tested

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Exhaled acetate | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled propionate | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled butyrate | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Flame ionization detector (GC- FID) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)

SECONDARY OUTCOMES:
Gut microbiota | within 4 days before the second test day
  Illumina sequencing of 16SrDNA and GC-FID
Fecal short-chain fatty acids | Within 4 days before the ingestion of chitin-glucan
  Gaz chromatography using Flame ionization detector (GC- FID)
Fecal conjugated-linoleic acids | Within 4 days before the ingestion of chitin-glucan
  Gaz chromatography using Flame ionization detector (GC- FID)
Fecal bile acids | Within 4 days before the ingestion of chitin-glucan
  Gas chromatography-mass spectrometry (GC/MS)
Gastro-intestinal symptom - discomfort | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - nausea | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - bloating | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - flatulences | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - gastrointestinal reflux | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - cramps | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - rumbling | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Gastro-intestinal symptom - burps | Before product ingestion (baseline) and 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 9 hours, 10 hours, 11 hours and 12 hours after product ingestion
  100 mm Visual analog scale (0 = no symptom, 100 = very severe symptom) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled C2 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled CO2 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled H2S | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled O2 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled N2 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled CH4 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled CO | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled H2 | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using Thermal Conductivity Detector (GC-TCD) - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)
Exhaled volatils compounds (for other short-chain fatty acids and other volatile organic compounds) | Before product ingestion (baseline) and 30 minutes, 2 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours and 12 hours after product ingestion
  Gaz chromatography using selected ion flow tube mass spectrometry - Area under the curve (calculated on 12 hours following product ingestion) - Comparison between the test day 0 (ingestion of maltodextrin) and the test day 2 (ingestion of chitin-glucan)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Delzenne, Prof, Principal Investigator — UCL
Locations (1):
- Center of Investigation in Clinical Nutrition, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared by the partners from the Consortium agreement.
  * exhaled volatile metabolites
  * gut microbiota derived metabolites
  * visual analog scales data
  * concomitant medication, inclusion/exclusion criteria, adverse event, food and beverages consummed.
  Data will be shared at the end of the study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At the end of the study
Access Criteria: Belonging to the project partener (Consortium agreement)

REFERENCES:
- [Derived] Neyrinck AM, Rodriguez J, Zhang Z, Seethaler B, Mailleux F, Vercammen J, Bindels LB, Cani PD, Nazare JA, Maquet V, Laville M, Bischoff SC, Walter J, Delzenne NM. Noninvasive monitoring of fibre fermentation in healthy volunteers by analyzing breath volatile metabolites: lessons from the FiberTAG intervention study. Gut Microbes. 2021 Jan-Dec;13(1):1-16. doi: 10.1080/19490976.2020.1862028. PMID 33461385